CLINICAL TRIAL: NCT02616159
Title: A Randomized, Controlled, Double-Blind Crossover Trial to Assess Effect of Oatmeal Varieties on Glycemic and Insulinemic Responses in Healthy Individuals
Brief Title: Effect of Oatmeal Varieties on Glycemic and Insulinemic Responses in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PEP-1519
Record Dates: First submitted 2015-11-24; First posted 2015-11-26 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2015-11

CONDITIONS: Glycemic Response

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Oatmeal 1 (Experimental): 40 g cereal
  Interventions: Other: Oatmeal
- Oatmeal2 (Experimental): 40 g cereal
  Interventions: Other: Oatmeal
- Oatmeal 3 (Experimental): 40 g cereal
  Interventions: Other: Oatmeal
- Ready to eat cereal (Placebo Comparator): 32.2 g cereal
  Interventions: Other: Oatmeal
- Hot cereal (Placebo Comparator): 28.8 g cereal
  Interventions: Other: Oatmeal

INTERVENTIONS:
Other: Oatmeal

SUMMARY:
The objectives of this study are to compare the glycemic and insulinemic responses over 3 hours elicited by 3 oatmeal varieties compared to each other and to controls of ready to eat and hot cereals.

DETAILED DESCRIPTION:
Participant eligibility will be screened at visit 1. The study will be a randomized, cross-over design. Participants will come to the study site on 5 separate occasions separated by a 2-day to 2-week washout period. Participants will arrive to the lab in a fasted state. 2 fasting blood samples will be collected, and further blood sampled will be taken over a 3-hour period post study product consumption.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant females, 18-75 years of age, inclusive
* Body mass index (BMI) ≥ 20.0 and < 35 kg/m² at screening (visit 1).
* Willing to maintain habitual diet, physical activity pattern, and body weight throughout the trial and to refrain from smoking for 12hr prior to each visit.
* Willing to maintain current dietary supplement use throughout the trial. On test days, subject agrees not to take any dietary supplements until dismissal from the GI labs. Failure to comply will result in a rescheduled test visit.
* Normal fasting serum glucose (<7.0mmol/L capillary corresponding to whole blood glucose <6.3mmol/L).
* Willing to abstain from alcohol consumption and avoid vigorous physical activity for 24 h prior to all test visits.
* Absence of health conditions that would prevent fulfillment of study requirements as judged by the Investigator on the basis of medical history.
* Understanding the study procedures and willing to provide informed consent to participate in the study and authorization to release relevant protected health information to the study investigator.

Exclusion Criteria:

* Failure to meet any one of the inclusion criteria
* Known history of AIDS, hepatitis, a history or presence of clinically important endocrine (including Type 1 or Type 2 diabetes mellitus), cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, biliary or GI disorders.
* Use of medications known to influence carbohydrate metabolism, including, but not limited to adrenergic blockers, diuretics, thiazolidinediones, metformin and systemic corticosteroids within 4 weeks of the screening visit, or with any condition which might, in the opinion of Dr. Wolever, the president of GI Testing, either: 1) make participation dangerous to the subject or to others, or 2) affect the results.
* Major trauma or surgical event within 3 months of screening.
* Unwillingness or inability to comply with the experimental procedures and to follow GI Labs safety guidelines.
* Known intolerance, sensitivity or allergy to any ingredients in the study products.
* Extreme dietary habits, as judged by the Investigator (i.e. Atkins diet, very high protein diets, etc).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
peak rise of blood glucose | 3 hours post dose

SECONDARY OUTCOMES:
Incremental area under the blood glucose and insulin response curves | 0-3 hours post dose
Peak rise of insulin | 0-3 hours post dose
Peak glucose and insulin concentrations | 0-3 hours post dose
Blood glucose and insulin concentrations at each time point over a 3hr period | 0-3 hours post dose

CONTACTS AND LOCATIONS:
Locations (1):
- Glycemic Index Laboratories, Toronto, Canada